CLINICAL TRIAL: NCT04280900
Title: Benefits of Therapy With Virtual Reality Exposure in the Treatment of Cocaine Use Disorders
Acronym: CORVI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: Fondation de l'Avenir, France (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RBHP 2019 BROUSSE; 2019-A02368-49 (Other: 2019-A02368-49)
Record Dates: First submitted 2020-02-18; First posted 2020-02-21 (Actual); Last update posted 2020-02-21 (Actual); Status verified 2020-02

CONDITIONS: Addiction; Cocaine-Related Disorders
Keywords: Cocaine-Related Disorders; Virtual Reality Exposure Therapy; Behavior Therapy
MeSH Terms: conditions — Behavior, Addictive; Cocaine-Related Disorders | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- cybertherapy (Experimental): use of cybertherapy (8 sessions) in addition to cognitive behavioral therapy (4 sessions) (pharmacological treatment are note modified)
  Interventions: Behavioral: Virtual Reality-Enhanced Cognitive Behavioral Therapy (VR-CBT); Behavioral: Treatment as usual
- Treatment as usual (Other): Treatment as usual is a cognitive behavioral therapy I (4 sessions) (pharmacological treatment are note modified)
  Interventions: Behavioral: Treatment as usual

INTERVENTIONS:
Behavioral: Virtual Reality-Enhanced Cognitive Behavioral Therapy (VR-CBT) — use of cybertherapy (8 sessions) in addition to cognitive behavioral therapy (4 sessions) (pharmacological treatment are note modified)
  Arms: cybertherapy
Behavioral: Treatment as usual — Treatment as usual is a cognitive behavioral therapy I (4 sessions) (pharmacological treatment are note modified)

SUMMARY:
Cocaine addiction is a multifactorial disease with important consequences: somatic, psychiatric... The number of applications for treatment for cocaine addiction is gradually increasing from year to year but no conventional treatment is available. New tools such as virtual reality could be used in this treatment. We propose to create a virtual reality program based on the analysis of high-risk relapse situations described by patients. We will then assess the effect of this cybertherapy on patients' relapse time and their desire to use cocaine

DETAILED DESCRIPTION:
In France, according to the Health Barometer 2017, cocaine testing has seen two decades of increases from 1.2% in 1995 to 5.6% in 2017, making it the second most widely used illicit substance. About 5% of cocaine users may become addicted in the first year of use, while 20% will develop long-term addiction. This dependence or substance use disorder is characterized in particular by a loss of control of cocaine use and continued use despite the negative consequences. Another of the central dimensions of this disorder is the craving (irresistible or irrepressible need or desire to consume) which is caused by internal or external stimuli. Craving is the cause of frequent loss of controls and re-consumption.

The treatment of cocaine addictions is generally based on a dual model of pharmacological treatment often aimed at limiting craving and psychotherapeutic treatment in order to alter the emotions and memory associated with cocaine use; for example: relearning product management when it comes to the subject.

In this context, the use of a 3D tool, which allows a gradual and well-detested exposure without confrontation, seems an interesting prospect. Virtual reality therapies have historically been known for treating phobias (fears). In addictions, exposure therapies are done in imagination and rarely with consumer-inducing situations. Since 2000, several researchers have successfully used virtual reality applications in addictions, but there is little data on objective assessments of the effectiveness of cybertherapy in the treatment of cocaine addictions.

All of these elements converge to propose a protocol called "CORVI" to evaluate the effectiveness of virtual reality exposure therapy as the management of patients with cocaine use disorder versus management classic.

The project is based on 3 phases: 1/construction of films that can be used in cybertherapy that reproduce situations in which there are stimuli generating "craving" to cocaine. 2/ Treatment of 2 randomized patient groups with and without cybertherapy (n-20/group) 3/Relapse evaluations at 1.2 and 3 months post-treatment

ELIGIBILITY:
Inclusion Criteria:

* suffering from a cocaine use disorder with craving criteria present according to the criteria of DSM 5
* wanting to stop cocaine use
* able to give informed consent to participate in research
* Covered by a Social Security plan.

Exclusion Criteria:

Patient with:

* psychiatric comorbidities (DSM 5) unstabilized
* dipsomaniac alcoholism
* an anteriority of one or more hypomanic or manic episodes
* unstabilized psychosis
* an unstabilized depression
* a severe suicidal risk
* a syndrome of dependence on products other than cocaine or tobacco
* unstabilized anxiety
* problems that hinder participation in 3D exposure, as a tendency to dissociation; phobias of the type of information (panic attacks and hypochondria...) severe dizziness...
* cognitive problems limiting or preventing the possibility of implementing coping or managing emotions or stimuli and disabilities to complete questionnaires
* a language barrier
* a serious intercurrent pathology
* the need for weekly individual follow-up Patient in a protected population such as pregnant women, lactating women, patients under guardianship, guardianship, deprived of freedoms, or in safeguarding justice

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-06-01 (Estimated); Primary Completion 2021-09-01 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of relapser patients at 3 months post-intervention | day 90 after intervention
  recovery in consumption of cocaine at M3 after intervention

SECONDARY OUTCOMES:
Craving score | day 30 after intervention
  evaluation of craving score (/10) compared to inclusion score
Craving score | day 90 after intervention
  evaluation of craving score (/10) compared to inclusion score
Score on the personal efficiency sentiment scale | day 30 after intervention
  Evaluation of the score on the personal efficiency sentiment scale
Score on the personal efficiency sentiment scale | day 90 after intervention
  Evaluation of the score on the personal efficiency sentiment scale
Consumption of quantity of cocaine | day 30 after intervention
  Evaluation of quantity of cocaine consumed
Consumption of quantity of cocaine | day 60 after intervention
  Evaluation of quantity of cocaine consumed
Consumption of quantity of cocaine | day 90 after intervention
  Evaluation of quantity of cocaine consumed
Frequency of consumption of cocaine | day 30 after intervention
  Evaluation of the frequency of cocaine consumption
Frequency of consumption of cocaine | day 60 after intervention
  Evaluation of the frequency of cocaine consumption
Frequency of consumption of cocaine | day 90 after intervention
  Evaluation of the frequency of cocaine consumption
Way of consumption of cocaine | day 30 after intervention
  Evaluation of the way of cocaine consumption
Way of consumption of cocaine | day 60 after intervention
  Evaluation of the way of cocaine consumption
Way of consumption of cocaine | day 90 after intervention
  Evaluation of the way of cocaine consumption
amount of cocaine consumed during relapse | day 30 after intervention
  Evaluation of cocaine amount consumed during relapse
amount of cocaine consumed during relapse | day 90 after intervention
  Evaluation of cocaine amount consumed during relapse
Frequence of cocaine consumed during relapse | day 30 after intervention
  Evaluation of cocaine frequence consumption during relapse
Frequence of cocaine consumed during relapse | day 90 after intervention
  Evaluation of cocaine frequence consumption during relapse
Percentage of relapser patients | day 30 after intervention
  recovery in relapser patients at M1 after intervention
Duration of abstinence | day 30 after intervention
  recovery of abstinence duration
Duration of abstinence | day 60 after intervention
  recovery of abstinence duration
Duration of abstinence | day 90 after intervention
  recovery of abstinence duration

CONTACTS AND LOCATIONS:
Overall Officials: Georges Brousse, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU Clermont Ferrand, Clermont-Ferrand, Auvergne, France